CLINICAL TRIAL: NCT05479864
Title: Single Level Anterior Cervical Corpectomy Without Posterior Stabilization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Ragab Hassan Alshemy, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: spine surgery
Record Dates: First submitted 2022-04-08; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Cervical Spine Fusion
MeSH Terms: conditions — Klippel-Feil Syndrome | interventions — Gene Fusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anterior cervical corpectomy and fusion (Other): removal of damaged vertebrae and intervertebral disc that are compressing the spinal cord and spinal nerves. Various graft materials or spacers are used to maintain height and stability followed by anterior plating
  Interventions: Procedure: anterior cervical corpectomy and fusion

INTERVENTIONS:
Procedure: anterior cervical corpectomy and fusion — removal of damaged vertebrae and intervertebral disc that are compressing the spinal cord and spinal nerves

SUMMARY:
evaluate and assess short term outcome of treating degenerative and non-degenerative cervical conditions with single level anterior cervical corpectomy without posterior fusion

DETAILED DESCRIPTION:
Cervical corpectomy is a procedure that removes damaged vertebrae and intervertebral disc that are compressing the spinal cord and spinal nerves. Various graft materials or spacers are used to maintain height and stability followed by anterior plating. It has an important role in the management of various degenerative, traumatic, neoplastic and infectious disorders of cervical spine.

While ACCF effectively decompresses the spinal cord, it is debated whether it can provide enough cervical stability, or an additional posterior fixation (PF) is required. Studies show that in multi-level anterior cervical corpectomy, additional posterior fixation provides extra support to improve cervical stability whether it is performed initially, or later as a supplementary surgery if material failure or instability occurred, On the other hand, in single level corpectomy, it remains controversial as single level ACCF showed sufficient stability in the majority of cases without additional support but pathologies affecting bone quality like infections and neoplasms seemed to be risk factor for construct failure and instability so additional PF was required .

ELIGIBILITY:
Inclusion Criteria:

- All patients with degenerative and non-degenerative cervical conditions (trauma, tumors and infections) treated with "single level anterior cervical corpectomy without posterior fusion

Exclusion Criteria:

* Patients who refuse to participate in the study
* Patients who are not available for 6 months follow up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Radiological parameter | Baseline
  * Bony fusion with no metal failure
  * presence of trabecular bridging and/or absence of motion

SECONDARY OUTCOMES:
Physiological parameter | baseline
  Percentage of improvement in NDI following surgical treatment during the follow up visits

REFERENCES:
- [Background] Nouri A, Tetreault L, Singh A, Karadimas SK, Fehlings MG. Degenerative Cervical Myelopathy: Epidemiology, Genetics, and Pathogenesis. Spine (Phila Pa 1976). 2015 Jun 15;40(12):E675-93. doi: 10.1097/BRS.0000000000000913. PMID 25839387
- [Background] Perez-Cruet MJ, Samartzis D, Fessler RG. Anterior cervical discectomy and corpectomy. Neurosurgery. 2006 Apr;58(4 Suppl 2):ONS-355-9; discussion ONS-359. doi: 10.1227/01.NEU.0000205285.20336.C2. PMID 16582660